CLINICAL TRIAL: NCT07254767
Title: Combination of Visuo-proprioceptive Virtual Walking and Neuromodulation to Reduce Neuropathic Pain in Individuals With Spinal Cord Injury
Brief Title: Virtual Walking and Neuromulation to Reduce Neuropathic Pain After a Spinal Cord Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Responsible Party: Principal Investigator, Cyril Duclos, Professor, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRIR-2025-2084
Record Dates: First submitted 2025-09-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; spinal cord injury; mixed methods; single subject design; tDCS; virtual reality; muscle vibration
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Single subject design with mixed methods
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3-Phase Arm (Experimental): Using repeated measurements over time, in three phases, i.e. an observation phase A, an intervention phase B and a post-intervention follow-up phase C, each participant will be his or her own control.
  Phase A : consists of an observational period without intervention, aimed at establishing a baseline and gaining a clearer understanding of the individual characteristics and patterns of neuropathic pain in each participant.
  Phase B : The intervention will be provided during Phase B. The intervention consists of starting neuromodulation 5min with tDCS alone, then adding virtual walking (virtual reality + corresponding somatosensory stimulation, via muscle vibration in the lower limbs) for the last 15min Phase C: follow up until 6monts post the end of the intervention.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS) combined with virtual reality and muscle vibration

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) combined with virtual reality and muscle vibration — tDCS will be delivered over the primary motor cortex (M1) to maximize the analgesic effect. The cathode will be positioned over the suborbital region, and the anode over M1 (position C3 or C4 of the international 10-20 system). A 2 mA direct current will be applied.
  Participants will observe, through virtual reality goggles (HTC Vive), an avatar walking from a first-person perspective, synchronized with the vibration pattern. Twelve vibrators will be placed transversely and bilaterally over the tendons of the main flexors and extensors of the lower limbs.
  The pattern used to trigger the vibrators is based on the natural sequence of gait movement. Muscle vibration induces a perception of movement in the direction of muscle elongation. The target frequency of the vibrators will be 80 Hz.
  The session will begin with 5 minutes of tDCS alone, and then for the last 15minutes the investigators will combine tDCS, virtual reality and muscle vibration.

SUMMARY:
The goal of this single-subject design is to evaluate an intervention combining neuromodulation, virtual reality, and muscle vibration to reduce neuropathic pain in individuals following a spinal cord injury.

The investigators aim to quantify the effects of the intervention on the intensity and characteristics of neuropathic pain, as well as its impact on daily functioning in individuals undergoing SCI rehabilitation. Additionally, the investigators seek to gain a better understanding of participants' experiences with the intervention by exploring effects not captured by standardized questionnaires, and by examining the role and meaning of the intervention in their management and experience of pain.

Finally, the investigators aim to assess the feasibility and clinical relevance of implementing this intervention in a rehabilitation setting.

All participants living with neuropathic pain following a spinal cord injury will take part in ten intervention sessions. They will also be invited to complete standardized questionnaires and participate in a semi-structured interview. In addition, their clinicians will be invited to participate in a focus group.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* a score of ≥ 4/10 on the Douleur Neuropathique en 4 Questions (DN4)
* classified AIS A to D
* neuropathic pain with an intensity of ≥ 4/10 on the simple numerical rating scale (This threshold is often chosen to better observe a potential analgesic effect)

Exclusion Criteria: The main exclusion criteria are contraindications to tDCS and virtual reality

* pregnancy,
* epilepsy,
* cancer,
* pacemaker,
* metallic implants in the brain or eyes,
* uncontrolled severe headaches,
* uncontrolled psychotic disorders,
* open scalp wounds,
* severe visual impairments. If participants have suffered a major traumatic brain injury with significant cognitive impairments, inclusion in the study will depend on the medical team's judgment. Finally, participants with allodynia in the areas where vibrators will be placed will not be included in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Phase A (baseline): once daily from Day 1 to Day 7 Phase B (intervention): before and after each session, 2-3 sessions per week, for up to 4 weeks (10 sessions total). Phase C (follow up): at 1 month and 4 months after the end of the intervention.
  Pain intensity will be measured with Numeric rating scale, an 11-point scale to measure pain intensity, ranging from 0 (no pain) to 10 (worst possible pain). In the case of pain after spinal cord injury, the minimum clinically significant change would be around 1.8 points. Test-retest reliability ranged from 0.63 to 0.92, with intra- and inter-rater reliability of 0.84-0.98

SECONDARY OUTCOMES:
Pain interference | Phase A (baseline): Day 1 and Day 7. Phase B (intervention): after session 5 (week 2) and session 10 (week 4). (10 sessions total, 2-3 per week, for up to 4 weeks) Phase C (follow up) : at 1 month and 4 months after the end of the intervention.
  The investigators extracted the interference section containing 3 items from the "international spinal cord injury pain basic data set data collection form - Version 3.0" in order to measure pain interference on daily activities, mood and sleep over the last 7 days. For each self-administered question, interference is measured on a scale from 0 (no interference) to 10 (maximum interference). The total score ranges from 0 to 30, a higher score means a greater pain interference.This questionnaire has been validated in people after spinal cord injury.
Pain characteristics | Phase A (baseline): Day 1 and Day 7. Phase B (intervention): after session 5 (week 2) and session 10 (week 4). (10 sessions total, 2-3 per week, for up to 4 weeks) Phase C (follow up): at 1 month and 4 months after the end of the intervention.
  Pain characteristics measured with PainDETECT. A tool initially developed to detect neuropathic components in people with chronic pain in the lumbar region. This questionnaire is increasingly used for other conditions, including post-spinal cord injury, helping to establish an individualized pain profile. It is also used in brain imaging studies. There are 9 items, 7 on sensory characteristics and 2 on temporal and spatial characteristics. It is scored from 0 to 38. A total of 19 or more indicates a high probability of having a neuropathic component.
Participant satisfaction rating for the Intervention | At the 10th (final) session (during phase B), in Week 4, assuming 10 sessions are conducted at a frequency of 2-3 per week.
  The research team developed a questionnaire to assess overall satisfaction with the intervention, as well as satisfaction with the timing, frequency, duration, content, and format of the sessions. There are 9 items, the satisfaction related to each item is scored on a scale 0 (not at all satisfied) to 10 (extremely satisfied). The total score ranges from 0 to 90, a higher score means a greater satisfaction of the participant regarding the intervention.
Qualitative themes from semi-structured interviews on perceived effects, embodiment, feasibility, and personal impact of the intervention in the participant with neuropathic pain after a spinal cord injury (SCI) | At the 10th (final) session (phase B), in week 4, assuming 10 sessions are conducted at a frequency of 2-3 per week
  Semi-structured interviews will be conducted with participants with neuropathic pain after a SCI. Each interview will last approximately 60 minutes and will follow a guide developed to structure the discussion. Thematic areas will include rehabilitation needs, overall experience with the intervention, perceived effects, embodiment, feasibility, suggestions regarding both positive and negative aspects, and for improving the intervention (for example in terms of effects or feasibility). How the intervention contributes to individuals' self-perception and interpretation of their pain experience will be also investigated. These interviews will be audio-recorded.
Qualitative themes identified through focus groups with clinicians on the perceived role, implementation, and impact of the intervention | 3 to 6months after the end of the intervention
  Focus group will be conducted with clinicians. Each interview will last approximately 90 minutes and will follow a guide developed to structure the discussion. Thematic areas will include the role of the intervention in patient care, clinical relevance, necessary changes and tools kit for implementation, perceived changes observed in patients, as well as both positive and negative aspects.
Intervention sessions adherence rate | At the end of phase B, in week 4, assuming 10 sessions are conducted at a frequency of 2-3 per week
  Adherence to intervention sessions will be collected. It will be calculated as a percentage: the number of sessions completed divided by the number of sessions planned, multiplied by 100. The total score ranges from 0% to 100%, with higher scores indicating greater adherence to the sessions.
Rate of submission of baseline questionnaires | When the participant has completed phase A. In phase A, the protocole includes 7 times of evaluation Day 1 to Day 7.
  The rate of submission of the evaluation questionnaires will be collected. It will be calculated as a percentage: the number of questionnaires completed divided by the number of questionnaires expected (phase A), multiplied by 100. The total score ranges from 0% to 100%, with higher scores indicating greater adherence to the questionnaire.
Recruitment rate | At the end of the project, after all participants have been recruited (in 2 years).
  The investigators will calculate the recruitment rate as the percentage of participants who actually enrolled in the study out of the total number of potential participants who were approached and expressed interest,multiplied by 100. The total score ranges from 0% to 100%, with higher scores indicating greater recruitment rate.
participants' perception of walking during the session | During phase B (intervention): after each intervention session, 2-3 sessions per week, for up to 4 weeks (10 sessions total)
  After each intervention session, the investigators will ask participants to rate their perception of walking during the intervention stimulation using a numeric rating scale between 0 "The perception was not at all a perception of gait motion" and 10 "The perception was definitely a perception of gait motion". If the score is below 5/10, open-ended questions such as "What did you feel during the sessions?" and "How would you describe your sensations?" to explore whether participants experienced a perception of walking, and to rate how strong that perception was on a scale from 0 to 10.
The session duration with the technologies (both installation and treatment) | During phase B (intervention): for each session, 2-3 sessions per week, for up to 4 weeks (10 sessions total)
  The total session duration, including the time required for installation and the actual treatment using the technologies, will be documented. Based on preliminary trials with partner patients, investigators expect an average duration of 40 minutes (20 minutes for installation and 20 minutes for treatment). Any deviations from this expected duration, including delays, will be documented and used to assess the feasibility of the project.

IPD SHARING:
Plan to Share IPD: Yes
Individual quantitative data will be included in the articles reporting the results of the study.

REFERENCES:
- [Background] Austin PD, Craig A, Middleton JW, Tran Y, Costa DSJ, Wrigley PJ, Siddall PJ. The short-term effects of head-mounted virtual-reality on neuropathic pain intensity in people with spinal cord injury pain: a randomised cross-over pilot study. Spinal Cord. 2021 Jul;59(7):738-746. doi: 10.1038/s41393-020-00569-2. Epub 2020 Oct 19. PMID 33077900
- [Background] Burke D, Fullen BM, Stokes D, Lennon O. Neuropathic pain prevalence following spinal cord injury: A systematic review and meta-analysis. Eur J Pain. 2017 Jan;21(1):29-44. doi: 10.1002/ejp.905. Epub 2016 Jun 24. PMID 27341614
- [Background] Chi B, Chau B, Yeo E, Ta P. Virtual reality for spinal cord injury-associated neuropathic pain: Systematic review. Ann Phys Rehabil Med. 2019 Jan;62(1):49-57. doi: 10.1016/j.rehab.2018.09.006. Epub 2018 Oct 9. PMID 30312665
- [Background] Widerstrom-Noga E, Biering-Sorensen F, Bryce T, Cardenas DD, Finnerup NB, Jensen MP, Richards JS, Siddall PJ. The international spinal cord injury pain basic data set. Spinal Cord. 2008 Dec;46(12):818-23. doi: 10.1038/sc.2008.64. Epub 2008 Jun 3. PMID 18521092
- [Background] Ummels D, Cnockaert E, Timmers I, den Hollander M, Smeets R. Use of Virtual Reality in Interdisciplinary Multimodal Pain Treatment With Insights From Health Care Professionals and Patients: Action Research Study. JMIR Rehabil Assist Technol. 2023 Nov 10;10:e47541. doi: 10.2196/47541. PMID 37948109
- [Background] Tapin A, Duclos NC, Jamal K, Duclos C. Perception of gait motion during multiple lower-limb vibrations in young healthy individuals: a pilot study. Exp Brain Res. 2021 Nov;239(11):3267-3276. doi: 10.1007/s00221-021-06199-1. Epub 2021 Aug 31. PMID 34463827
- [Background] Sreeraj VS, Arumugham SS, Venkatasubramanian G. Clinical Practice Guidelines for the Use of Transcranial Direct Current Stimulation in Psychiatry. Indian J Psychiatry. 2023 Feb;65(2):289-296. doi: 10.4103/indianjpsychiatry.indianjpsychiatry_496_22. Epub 2023 Jan 30. No abstract available. PMID 37063621
- [Background] Matamala-Gomez M, Donegan T, Bottiroli S, Sandrini G, Sanchez-Vives MV, Tassorelli C. Immersive Virtual Reality and Virtual Embodiment for Pain Relief. Front Hum Neurosci. 2019 Aug 21;13:279. doi: 10.3389/fnhum.2019.00279. eCollection 2019. PMID 31551731
- [Background] Luo L, Liu Y, Huang L, Ming Z, Cao J. Neuropathic Pain Experience and Self-Management Strategies of Spinal Cord Injury Patients: A Meta-Synthesis of Qualitative Studies. Pain Manag Nurs. 2025 Jul 26:S1524-9042(25)00215-2. doi: 10.1016/j.pmn.2025.06.015. Online ahead of print. PMID 40716978
- [Background] Loh E, Mirkowski M, Agudelo AR, Allison DJ, Benton B, Bryce TN, Guilcher S, Jeji T, Kras-Dupuis A, Kreutzwiser D, Lanizi O, Lee-Tai-Fuy G, Middleton JW, Moulin DE, O'Connell C, Orenczuk S, Potter P, Short C, Teasell R, Townson A, Widerstrom-Noga E, Wolfe DL, Xia N, Mehta S. The CanPain SCI clinical practice guidelines for rehabilitation management of neuropathic pain after spinal cord injury: 2021 update. Spinal Cord. 2022 Jun;60(6):548-566. doi: 10.1038/s41393-021-00744-z. Epub 2022 Feb 5. PMID 35124700
- [Background] Li C, Jirachaipitak S, Wrigley P, Xu H, Euasobhon P. Transcranial direct current stimulation for spinal cord injury-associated neuropathic pain. Korean J Pain. 2021 Apr 1;34(2):156-164. doi: 10.3344/kjp.2021.34.2.156. PMID 33785667
- [Background] Leemhuis E, Esposito RM, De Gennaro L, Pazzaglia M. Go Virtual to Get Real: Virtual Reality as a Resource for Spinal Cord Treatment. Int J Environ Res Public Health. 2021 Feb 13;18(4):1819. doi: 10.3390/ijerph18041819. PMID 33668438
- [Background] Le Franc S, Bonan I, Fleury M, Butet S, Barillot C, Lecuyer A, Cogne M. Visual feedback improves movement illusions induced by tendon vibration after chronic stroke. J Neuroeng Rehabil. 2021 Oct 30;18(1):156. doi: 10.1186/s12984-021-00948-7. PMID 34717672
- [Background] Labbe, D. R., Kouakoua, K., Aissaoui, R., Nadeau, S., & Duclos, C. (2021). Proprioceptive Stimulation Added to a Walking Self-Avatar Enhances the Illusory Perception of Walking in Static Participants. Frontiers in Virtual Reality, 2. https://www.frontiersin.org/article/10.3389/frvir.2021.557783
- [Background] Krasny-Pacini A, Evans J. Single-case experimental designs to assess intervention effectiveness in rehabilitation: A practical guide. Ann Phys Rehabil Med. 2018 May;61(3):164-179. doi: 10.1016/j.rehab.2017.12.002. Epub 2017 Dec 15. PMID 29253607
- [Background] Jutzeler CR, Huber E, Callaghan MF, Luechinger R, Curt A, Kramer JL, Freund P. Association of pain and CNS structural changes after spinal cord injury. Sci Rep. 2016 Jan 6;6:18534. doi: 10.1038/srep18534. PMID 26732942
- [Background] Imai R, Osumi M, Morioka S. Influence of illusory kinesthesia by vibratory tendon stimulation on acute pain after surgery for distal radius fractures: a quasi-randomized controlled study. Clin Rehabil. 2016 Jun;30(6):594-603. doi: 10.1177/0269215515593610. Epub 2015 Jul 21. PMID 26198893
- [Background] Hallstrom H, Norrbrink C. Screening tools for neuropathic pain: can they be of use in individuals with spinal cord injury? Pain. 2011 Apr;152(4):772-779. doi: 10.1016/j.pain.2010.11.019. Epub 2011 Jan 26. PMID 21272997
- [Background] Gupta A, Scott K, Dukewich M. Innovative Technology Using Virtual Reality in the Treatment of Pain: Does It Reduce Pain via Distraction, or Is There More to It? Pain Med. 2018 Jan 1;19(1):151-159. doi: 10.1093/pm/pnx109. PMID 29025113
- [Background] Freynhagen R, Tolle TR, Gockel U, Baron R. The painDETECT project - far more than a screening tool on neuropathic pain. Curr Med Res Opin. 2016 Jun;32(6):1033-57. doi: 10.1185/03007995.2016.1157460. Epub 2016 Mar 11. PMID 26907456
- [Background] Finnerup NB. Neuropathic pain and spasticity: intricate consequences of spinal cord injury. Spinal Cord. 2017 Dec;55(12):1046-1050. doi: 10.1038/sc.2017.70. Epub 2017 Jul 11. PMID 28695904
- [Background] Duclos C, Kemlin C, Lazert D, Gagnon D, Dyer JO, Forget R. Complex muscle vibration patterns to induce gait-like lower-limb movements: proof of concept. J Rehabil Res Dev. 2014;51(2):245-51. doi: 10.1682/JRRD.2013.04.0079. PMID 24933722
- [Background] Austin PD, Siddall PJ. Virtual reality for the treatment of neuropathic pain in people with spinal cord injuries: A scoping review. J Spinal Cord Med. 2021 Jan;44(1):8-18. doi: 10.1080/10790268.2019.1575554. Epub 2019 Feb 1. PMID 30707649